CLINICAL TRIAL: NCT04645576
Title: Evaluation of the Efficacy and Safety of an Injectable Hyaluronic Acid-based Filler, Art Filler® Volume: Comparative Single-blind Study of the Non-inferiority Versus Juvéderm® Voluma on the Midface, Temple and Jaw-line and Non-comparative Study on the Chin
Brief Title: Evaluation of the Efficacy and Safety of an Injectable Hyaluronic Acid-based Filler, Art Filler® Volume: Comparative Single-blind Study of the Non-inferiority Versus Juvéderm® Voluma on the Midface, Temple and Jaw-line and Non-comparative Study on the Chin. (AF3)
Acronym: AF3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires FILLMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF3:2018-A00287-48; 2018-A00287-48 (Other: ANSM)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: During the period of this clinical trial (18 months), only two products will be used for the aesthetic procedures (Art Filler Volume and Juvéderm Voluma).
  This prospective study will analyze 120 patients maximum who will receive dermal filler injections to the midface, temple, chin and jaw-line (cross-injection is authorized with maximum 2 zones per subject). The injections will be administered in a randomly assigned split-face design, except for the chin. One side of the subject's face will receive Art Filler Volume according to the randomization table, whereas the other side will receive Juvéderm Voluma injections in a blinded manner for the subjects (single blinded). The chin will only receive one injection of Art Filler Volume.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Midface zone (Other): Injection in the mid-facial areas (split-face). One side of the subject's face will receive Art Filler Volume according to the randomization table, whereas the other side will receive Juvéderm Voluma injections in a blinded manner for the subjects (single blinded).
  Interventions: Device: Face correction with injectable fillers
- Temple (Other): Injection in the temples (split-face). One side of the subject's face will receive Art Filler Volume according to the randomization table, whereas the other side will receive Juvéderm Voluma injections in a blinded manner for the subjects (single blinded).
  Interventions: Device: Face correction with injectable fillers
- Jaw-line (Other): Injection in the jaw-line areas (split-face). One side of the subject's face will receive Art Filler Volume according to the randomization table, whereas the other side will receive Juvéderm Voluma injections in a blinded manner for the subjects (single blinded).
  Interventions: Device: Face correction with injectable fillers
- Chin (Experimental): The chin will only receive one injection of Art Filler Volume.
  Interventions: Device: Face correction with injectable fillers

INTERVENTIONS:
Device: Face correction with injectable fillers — Injection of hyaluronic acid-based fillers

SUMMARY:
The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume. These fillers (also known as soft tissue augmentation devices) can restore the age-related volume loss of the face, balance the disproportions or correct topographical anomalies. A previous study has already shown the efficacy of Art Filler Volume on the midface, but this study was not comparative. It was thus interesting to compare the efficacy of Art Filler Volume to a reference product but also to test its efficacy on other areas including the temple, jaw-line and chin.

DETAILED DESCRIPTION:
The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume. These fillers (also known as soft tissue augmentation devices) can restore the age-related volume loss of the face, balance the disproportions or correct topographical anomalies. A previous study has already shown the efficacy of Art Filler Volume on the midface, but this study was not comparative. It was thus interesting to compare the efficacy of Art Filler Volume to a reference product but also to test its efficacy on other areas including the temple, jaw-line and chin.

In this context, it is proposed to conduct, in post-CE marking, a randomized, prospective and comparative study in order to document, an adequate aesthetic correction of the treated areas as well as their immediate and long-term tolerance. This study aims to document the filling capacity of Art Filler Volume, in relation to a product technically of the same order and considered as a reference2,3,4,5 (this study will be comparative on temple / midface and jawline but no on the chin were only Art Filler Volume will be injected). To do this, subjects in whom a correction of mid-facial areas and / or temple and / or jaw-lines and / or chin is sought, will be included. The aesthetic correction will be appreciated at 3 weeks. Subjects will be followed over 18 months. The persistence of the correction will be evaluated at 3, 6, 9, 12, 15 and 18 months.

No corrective injections with the products under study will be allowed. Each subject could be injected for maximum 2 different zones.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who had signed a written informed consent
2. Man or Woman with an age ≥ 19 years old
3. Subject having a Fitzpatrick Phototype I to IV (annex 6)
4. Subject having a score of ≥ 2 in Global aesthetic 6-point scale scoring system on at least one area of interest (chin, midface, temples or jaw lines) (annex 1.1)
5. Subject having at least one of the following scales by clinical scoring (annex 1.2/1.3/1.4/1.5)

   * a grade of 2 or 3 on the ACRS Scale
   * a grade of 2 or 3 score on the MMVS Scale
   * a grade of 2 or 3 or 4 score on ATHS Scale
   * a grade of 2 or 3 score with NCJLS Scale
6. Subject registered with health insurance regimen
7. Woman agreeing to take a pregnancy test

Exclusion Criteria:

1. Subject currently participating in another clinical study related to pharmaceuticals or medical devices or being in exclusion period of another clinical study.
2. Subject deprived of freedom by an administrative or legal decision
3. Subject who have received indemnification of 4500 € during the 12 previous months for his/her participation in clinical trials (including his participation in this study).
4. Subject who had facial injections/implants of any non-absorbable fillers in her/his whole life.
5. Subject who had laser sessions for skin rejuvenation or a laser resurfacing during the 12 previous months or a surgical facelift during the 2 years before the study.
6. Subject with a history of facial aesthetic injection (hyaluronic acid within the previous year, botulinum toxin within the last 6 months and long-term temporary injectable implants (semi-permanent implants) within the previous 2 years).
7. Subject with a skin-retaining device on the face (mesh, gold wire, liquid silicone or other particulate material).
8. Subject who undergo a non-invasive rejuvenation method such as moderate to deep peeling, ultrasound, radiofrequency devices or lasers within the last 6 months.
9. Subject with a history of severe multiple allergies or anaphylactic shock.
10. Subject with a known hypersensitivity to hyaluronic acid, Lidocaine and/or other components of Art Filler® Volume and Juvéderm Voluma solutions.
11. Subject with a known hypersensitivity to chlorhexidine.
12. Subject with a known hypersensitivity to lidocaine or local amide anesthetics.
13. Subject tending to develop inflammatory skin diseases or hypertrophic scars.
14. Subject with a history of streptococcal disease (recurring angina, rheumatic fever).
15. Subject with oral or injectable corticoid treatment (or not stopped for at least 3 months). Inhaled corticoids are permitted as well as topical corticotherapy not involving the head or the neck.
16. Subjects with any concomitant treatment (or not stopped for at least a year) by immunosuppressant or chemotherapy.
17. Subject with a history of radiotherapy involving the head and the neck within the previous year.
18. Subject with a history or a disease associated to the autoimmune or connective tissue disease.
19. Subject presenting at his/her face and/or neck any skin disease, or an acute inflammatory reaction or a bacterial/viral infection or who had such an episode within the previous 6 weeks.
20. Subject who took aspirin or anticoagulants at regular doses in the last 15 days prior to the act.
21. Subject who has permanently been exposed to the sun or the UV during the last 15 days.
22. Subject with dermatological condition or inflammation on or near the area to be treated (according to the opinion of the investigator).
23. Pregnant or lactating woman.
24. Subject with epilepsy not controlled by treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Volume correction on D21 with Art Filler Volume product | D21 (21 days after the injections)
  Objectively measure after a single injection of Art Filler® Volume the restoration of the chin volume versus a reference product, Juvéderm® Voluma, the restoration of midface, temple, and jaw-line from volumes baseline (D0) to D21 according to a global Aesthetic 6-point scale clinical scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Ferial FANIAN, MD, Study Director — Laboratoires FILLMED
Locations (1):
- Dr Frédéric Braccini, Nice, France

IPD SHARING:
Plan to Share IPD: No